CLINICAL TRIAL: NCT04301284
Title: Phase 2 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of CAD-1883 in Adults With Spinocerebellar Ataxia (Synchrony-1)
Brief Title: Study of CAD-1883 for Spinocerebellar Ataxia
Acronym: Synchrony-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In January 2021 Novartis acquired Cadent Therapeutics. As part of a pipeline reassessment, the Synchrony-1 trial will not proceed as initially scheduled.
Sponsor: Cadent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAD1883-211
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Spinocerebellar Ataxias; Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia Type 3; Spinocerebellar Ataxia Type 6; Spinocerebellar Ataxia Type 7; Spinocerebellar Ataxia Type 8; Spinocerebellar Ataxia Type 10; Spinocerebellar Ataxia Type 17; ARCA1 - Autosomal Recessive Cerebellar Ataxia Type 1
Keywords: Ataxia; SCA
MeSH Terms: conditions — Spinocerebellar Ataxias; Machado-Joseph Disease; Spinocerebellar ataxia 8; Spinocerebellar Ataxia 10; Olivopontocerebellar Atrophy V; Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAD-1883 (Experimental): Capsules of 150 mg of CAD-1883 will be administered orally, twice daily (BID). The second daily dose will be taken 8 hours (+/- 2 hours) after the first daily dose.
  The initial dose regimen evaluated will be 150 mg BID. Additional dose regimens up to 600 mg BID will be determined based on forthcoming clinical data.
  Interventions: Drug: CAD-1883
- Placebo (Placebo Comparator): Matching placebo will be provided in capsules, to be administered orally, twice daily. The second daily dose will be taken 8 hours (+/- 2 hours) after the first daily dose.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CAD-1883 — 150 mg filled capsules
  Arms: CAD-1883
Drug: Placebos — capsules
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 2 study evaluating oral administration of CAD-1883 in the treatment of adults with a genotypic diagnosis of Spinocerebellar Ataxia (SCA). This study offers the opportunity to understand the safety, tolerability, and efficacy of CAD-1883 in the SCA patient population.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 2 study evaluating oral administration of CAD-1883 in the treatment of adults with a genotypic diagnosis of SCA using multiple dose levels. The study will include multiple cohorts of 16 patients each where 12 patients will be randomized to CAD-1883 and 4 to matching placebo.

Potential subjects will undergo a screening period (14 to 28 days), a baseline (Day 1) visit, and a 12-week treatment period. A follow-up visit will occur 4 weeks after the end of the treatment period. The total duration of individual subject participation may be up to 20 weeks, depending on the duration of the screening period.

The study will assess safety by adverse events, vital signs, laboratory parameters (including chemistry, hematology and urinalysis); pharmacokinetics of CAD-1883; and efficacy measures by Scale for the Assessment and Rating of Ataxia (SARA), clinician/patient rating of ataxia and symptoms, patient quality of life measures and wearable sensors to capture falls and gait measurements.

For planning purposes, the anticipated study completion date assumes evaluation of 3 cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Prior Spinocerebellar Ataxia (SCA) diagnosis of the following SCA genotypes: SCA1, 2, 3, 6, 7, 8, 10, 17, or Autosomal Recessive Cerebellar Ataxia Type 1 (ARCA1).
* Scale for the Assessment and Rating of Ataxia (SARA) Total score ≥8 and <30 at Screening
* SARA item #1 (gait) score of ≥2 at Screening
* Ability to ambulate 8 meters at Screening without assistance from another person

Key Exclusion Criteria:

* Neurological condition other than SCA that could predominantly explain or contribute significantly to the subjects' symptoms of ataxia or that could confound the assessment of ataxia symptoms (e.g., chronic alcoholism, vitamin deficiencies, multiple sclerosis, Parkinson's disease, Friedreich's ataxia, vascular disease, tumors, paraneoplastic disease, head injury, idiopathic late onset ataxia, multisystem atrophy, stroke, arthritis, cerebral palsy, spasticity of unknown origin).
* Moderate or severe scores on the following Inventory of Non-Ataxia Signs (INAS) items at Screening: Dystonia: at least 3 of 5 items; Spasticity: at least 2 of 3 items; Rigidity: at least 2 of 3 items

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of oral administration of CAD-1883 versus placebo: Incidence of Adverse Events | 12 week treatment period
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Collaborative Neuroscience Network, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida: Ataxia Research Center, Tampa, Florida
  - Houston Methodist Research Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: No